CLINICAL TRIAL: NCT03190330
Title: A Prospective, Multicenter, Open Label Single Arm Phase IV Clinical Trial to Assess Safety of ImbruvicaTM (Ibrutinib Capsules 140 mg) in Indian Patients With Chronic Lymphocytic Leukemia or Mantle Cell Lymphoma Who Have Received at Least One Prior Therapy or Chronic Lymphocytic Leukemia With 17p Deletion
Brief Title: A Study to Assess Safety of ImbruvicaTM in Indian Participants With Chronic Lymphocytic Leukemia or Mantle Cell Lymphoma Who Have Received at Least One Prior Therapy or Chronic Lymphocytic Leukemia With 17p Deletion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Private Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108316; 54179060LYM4005 (Other: Johnson & Johnson Private Limited)
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ibrutinib (Experimental): Participants will receive ibrutinib 420 milligram (mg) (three 140 mg capsules) as a single daily dose for chronic lymphocytic leukemia (CLL) and 560 mg (four 140 mg capsules) as a single daily dose for mantle cell lymphoma (MCL) for up to 12 months or till disease progression, whichever is earlier.
  Interventions: Drug: Ibrutinib 420 mg; Drug: Ibrutinib 560 mg

INTERVENTIONS:
Drug: Ibrutinib 420 mg — Ibrutinib capsule administered orally at a dose of 420 mg for CLL participants.
  Other Names: Imbruvica
Drug: Ibrutinib 560 mg — Ibrutinib capsule administered orally at a dose of 560 mg for MCL participants.
  Other Names: Imbruvica

SUMMARY:
The primary purpose of this study is to evaluate the post-marketing safety of ImbruvicaTM (ibrutinib capsule 140 milligram [mg]) under actual conditions of use, and to understand the incidence of adverse events (AEs) (serious and non-serious AEs).

ELIGIBILITY:
Inclusion Criteria:

* Chronic lymphocytic leukemia (CLL) or mantle cell lymphoma (MCL) participants being newly initiated on Imbruvica treatment (ibrutinib capsule 140 milligram [mg]) based on independent clinical judgment of treating physicians as per locally approved prescribing information
* Must give a written informed consent indicating that they understand the purpose and are willing to participate in the study and allowing data collection and source data verification in accordance with regulatory requirements

Exclusion Criteria:

* Participants who are not eligible to receive Imbruvica as per the locally approved prescribing information
* Participants participating or planning to participate in any interventional drug trial during the course of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Private Limited Clinical Trial, Study Director — Johnson & Johnson Private Limited
Locations (10):
- India (10):
  - Avron Hospitals Pvt. Ltd, Ahmedabad
  - Post Graduate Institute of Medical Education And Research PGIMER, Chandigarh
  - Basavatarakam Indo-American Hospital, Hyderabad
  - Bhagwan Mahaveer Cancer Hospital & Research Centre, Jaipur
  - Cytecare Hospitals Pvt. Ltd, Karnataka
  - Apollo Multispeciality Hospital Ltd, Kolkata
  - Tata Medical Center, Kolkata
  - Jawaharlal Institute of Postgraduate Medical Education and Research, Puducherry
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
  - Noble Hospital Pvt Ltd, Pune

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Since the aim of the study was to assess the safety of Imbruvica (Ibrutinib 140 milligrams [mg]), combined data of enrolled participants with either chronic lymphocytic leukemia (CLL) or mantle cell lymphoma (MCL) was collected and analyzed as planned in the protocol.
Groups:
- Ibrutinib: Enrolled participants were prescribed ibrutinib as per locally approved prescribing information: a single daily dose of ibrutinib 420 mg (3 capsules of 140 mg) for participants with CLL and ibrutinib 560 mg (4 capsules of 140 mg) for participants with MCL, for up to 12 months or till disease progression, whichever was earlier.
Period: Overall Study
Arm/Group | Ibrutinib
Started | 75
Participants With CLL | 67
Participants With MCL | 8
Completed | 55
Not Completed | 20
Not completed — Adverse Event | 2
Not completed — Death | 10
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 6
Not completed — Progressive Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 75
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  India | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Any AE occurred at or after the initial administration of study drug up to maximum of 30 days after last dose was considered as treatment emergent.
Time Frame: Day 1 up to 30 days after last dose of study drug (up to 13 months)
Population: Safety analysis set included all participants who had signed the informed consent form (ICF) and received at least one dose of ibrutinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib
Number analyzed (Participants) | 75
Participants | 62

2. Primary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was an AE which resulted in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Any AE occurred at or after the initial administration of study drug up to maximum of 30 days after last dose was considered as treatment emergent.
Time Frame: Day 1 up to 30 days after last dose of study drug (up to 13 months)
Population: Safety analysis set included all participants who had signed the ICF and received at least one dose of ibrutinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib
Number analyzed (Participants) | 75
Participants | 23

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days after last dose of study drug (up to 13 months)
Description: Safety analysis set included all participants who had signed the ICF and received at least one dose of ibrutinib.
Arm/Group | Ibrutinib
All-Cause Mortality (participants affected / at risk) | 10/75
Serious Adverse Events (participants affected / at risk) | 23/75
Other Adverse Events (participants affected / at risk) | 55/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib (N=75)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Acute Coronary Syndrome (Cardiac disorders) | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Disease Progression (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Pyrexia (General disorders) | 4
Hepatic Function Abnormal (Hepatobiliary disorders) | 1
Brain Abscess (Infections and infestations) | 1
Bronchopulmonary Aspergillosis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cerebral Aspergillosis (Infections and infestations) | 1
Covid-19 (Infections and infestations) | 3
Oral Candidiasis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis Fungal (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib (N=75)
Anaemia (Blood and lymphatic system disorders) | 12
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 4
Vertigo (Ear and labyrinth disorders) | 4
Conjunctival Haemorrhage (Eye disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 2
Mouth Ulceration (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 7
Mucosal Inflammation (General disorders) | 2
Non-Cardiac Chest Pain (General disorders) | 2
Pain (General disorders) | 2
Pyrexia (General disorders) | 8
Covid-19 (Infections and infestations) | 3
Furuncle (Infections and infestations) | 5
Pneumonia (Infections and infestations) | 4
Urinary Tract Infection (Infections and infestations) | 4
Decreased Appetite (Metabolism and nutrition disorders) | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 7
Neuropathy Peripheral (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2
Blister (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2022-10-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT03190330/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT03190330/SAP_001.pdf